CLINICAL TRIAL: NCT06598761
Title: Postoperative Adjuvant Immunotherapy Combined with Radiotherapy Versus Surgery Alone in Locally Advanced Upper Tract Urothelial Carcinoma: a Prospective Observational Cohort Study
Brief Title: Postoperative Adjuvant Immunotherapy Combined with Radiotherapy Versus Surgery Alone in Locally Advanced UTUC
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, LI xiaoying, Vice Director of the Department of Radiation Oncology, Peking University First Hospital
Other Study IDs: LUXUS 2.1
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Ureter Cancer; Renal Pelvic Carcinoma; Advanced Urothelial Carcinoma
Keywords: upper tract urothelial carcinoma; Radiotherapy; Immunotherapy; Combined therapy; Prospective cohort study
MeSH Terms: conditions — Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observation cohort: Patients in the observation group were T3-4 or N+ UTUC patients who were intolerant to chemotherapy or refused chemotherapy after radical surgery. No postoperative treatment was performed, and the patients were regularly rechecked.
  Interventions: Other: surveillance alone
- Postoperative immunotherapy+radiotherapy: Adjuvant Immunotherapy: Immunotherapy drug of choice is tirilizumab, which has received national recommendations in metastatic uroepithelial cancer. Tirelizumab 200mg Q3w; the duration of immunotherapy is recommended for at least 1 year.
  Adjuvant radiotherapy can be given concurrently or sequentially with adjuvant immunotherapy; it is recommended that radiotherapy can be started within 4-6 weeks after surgery. Rotational intensity-modulated radiotherapy (VMAT), daily image-guided radiotherapy (Daily IGRT) techniques are used.
  Interventions: Combination Product: Immunotherapy+radiotherapy

INTERVENTIONS:
Combination Product: Immunotherapy+radiotherapy — Adjuvant Immunotherapy: Immunotherapy drug of choice is tirilizumab, which has received national recommendations in metastatic uroepithelial cancer. Tirelizumab 200mg Q3w; the duration of immunotherapy is recommended for at least 1 year.
  Adjuvant radiotherapy can be given concurrently or sequentially with adjuvant immunotherapy; it is recommended that radiotherapy can be started within 4-6 weeks after surgery. Rotational intensity-modulated radiotherapy (VMAT), daily image-guided radiotherapy (Daily IGRT) techniques are used.
  Groups: Postoperative immunotherapy+radiotherapy
Other: surveillance alone — Patients recieve surveillance alone without any adjuvant interventions until any disease progression endpoints occur.
  Groups: Observation cohort

SUMMARY:
This is a prospective cohort study to analyse the safety and efficacy of postoperative adjuvant radiotherapy combined with immunotherapy versus surgery alone group of UTUC patients with T3-4 stages or lymph nodes metastasis(N+) status.

DETAILED DESCRIPTION:
This study is a prospective cohort study.

1. Observation group: patients in the observation group were T3-4,N+ pyeloureteral cancer patients who did not tolerate chemotherapy or refused chemotherapy after radical surgery. No treatment will be given after surgery, and regular review will be conducted.
2. Postoperative immunotherapy+radiotherapy group:

Adjuvant immunotherapy: the immunotherapy drug choice is tirilizumab, which has been recommended in metastatic uroepithelial cancer in China. Tirelizumab 200mg Q3w; the duration of immunotherapy is recommended to be used for at least 1 year.

Adjuvant radiotherapy can be given concurrently or sequentially with adjuvant immunotherapy; it is recommended that radiotherapy can be started within 4-6 weeks after surgery. Rotational intensity-modulated radiotherapy (VMAT), daily image-guided radiotherapy (Daily IGRT) technique is used.

Irradiation range:

Renal pelvis and upper ureter: ipsilateral renal fossa, para-abdominal aorta (including upper ureteral alignment area), common iliac lymph node area; Middle and lower ureteral carcinoma: parabasal abdominal aorta (renal hilar vessels and following levels), common iliac lymph node area (right side needs to include paraventricular lymph node area) + internal and external iliac lymph node area + middle and lower ureteral alignment area, entrance of the ureteral bladder.

Radiotherapy dose: 45-50Gy/25f/5w, 62.5Gy/25f/5w regimen was given to suspected metastatic lymph nodes visible on imaging. Ensure that normal tissue is within the dose limits.

Note: The right tumour para-abdominal aortic lymph node drainage area needs to include: para vena cava + intervening vena cava + left para-abdominal aorta Left tumour para-abdominal lymph node drainage area needs to include: intervening vena cava + left para-abdominal aorta

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients after radical nephroureterectomy with full-length nephroureterectomy and pathologically confirmed cancer of the renal pelvis or ureter, AJCC staging (8th edition) containing one of the following factors: pT3-4, pN+; 2) Patients with creatinine eGFR <60 min/L. or underlying disease refusing to tolerate chemotherapy.

3)18≤age≤80 years old; 4)Completion of abdominopelvic CT 4 weeks prior to enrolment. 5)Except for cutaneous non-melanoma and ductal carcinoma in situ of the breast, the patient has not suffered from any other malignant disease within the last 5 years; 6)Willing to participate in perfecting the necessary examinations and follow-up visits for the sake of the study, and willing to provide written informed consent.

All of the above need to be fulfilled:

Expected survival > 6 months; KPS > 70 points; Leukocytes ≥ 3.5 x 109/l,Neutrophils ≥ 1.5 x 109/l, Platelets ≥ 100.0 x 109/l, Haemoglobin ≥ 90g/l.

Exclusion Criteria:

* 1) Distant metastases already found at the time of surgery; non-R0 resected patients 2) History of pelvic and abdominal radiotherapy; history of inflammatory bowel disease; history of systemic chemotherapy; (3) Pregnant or breastfeeding women; or women of childbearing potential who are not using reliable contraception; (4) History of malignant tumour (except skin cancer that is not malignant melanoma and cervical cancer in situ, tumours that have been cured for more than 5 years) 5) weight loss > 10% within 6 months 6) Presence of active infections in those with pre-existing or co-existing bleeding disorders 7) clinically significant cardiac disease (e.g., hypertension controlled by medication, unstable angina pectoris, New York Heart Association (NYHA) class ≥ II congestive heart failure, unstable symptomatic arrhythmia, or class ≥ II peripheral vascular disease); 8) Psychological, family, and social factors leading to lack of informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pT3-4/N+ UTUC patients who were eligible for enrolment and signed the informed consent could be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
DFS | 1-year and 3-year
  Disease-free survival，The time between the date of randomization and the date of first documented recurrence (local urothelial tract, local non-urothelial tract or distant), or death due to any cause, whichever occurs first.)

SECONDARY OUTCOMES:
OS | 1-year and 3-year
  overall survival，the time from randomization to the date of death from any cause
CSS | 1-year and 3-year
  Cancer-specific survival，the time from randomization to the date of death due to disease (urothelial cancer).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Departmeng of Urology, Peking University First Hospital, Beijing
  - Department of Radiotherapy Oncology, Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol